CLINICAL TRIAL: NCT02378909
Title: Diabetic Wound Healing and Its Relationship to Vascular Circulation.
Brief Title: Wound Healing Process in Diabetic Neuropathy and Diabetic Neuroischemia
Acronym: Geko
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manchester (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government); Firstkind Ltd (Industry)
Responsible Party: Principal Investigator, Ahmad Najib bin Hasan, Mr, University of Manchester
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: UManchester
Record Dates: First submitted 2015-02-26; First posted 2015-03-04 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Active Comparator): Diabetic Neuropathy with electrical stimulation device and standard of care.
  Interventions: Device: Electrical stimulation device.
- Group 2 (No Intervention): Diabetic neuropathy with standard of care.
- Group 3 (Active Comparator): Diabetic neuroischemia with electrical stimulation device and standard of care.
  Interventions: Device: Electrical stimulation device.
- Group 4 (No Intervention): Diabetic neuroischemia with standard of care.

INTERVENTIONS:
Device: Electrical stimulation device. — In the intervention group, all participants will receive Geko device which will produce electrical stimulation to enhance wound healing. This is the non- invasive device, self adhesive, light and does not restrict the patient's movement. Wound will be measured at the beginning of the study (before the device is applied) and after the study is complete. Blood and wound tissue samples will also be taken pre and post electrical stimulation to observe the effect of electrical stimulation on wound healing in people with diabetes.
  Other Names: GekoTM Device
  Arms: Group 1; Group 3

SUMMARY:
Diabetes mellitus is one of the leading causes of illness worldwide. Diabetes can affect nerves, skin and blood vessels. Diabetics with problems in their nerves can lose the sense of touch in their feet (called neuropathy) and so may unknowingly cause damage to the skin resulting in skin loss or an 'ulcer'. Diabetics also have difficulty healing any damaged tissues especially if the patients have diseased blood vessels causing a lack of blood to areas of the body including the feet (called ischaemia).

DETAILED DESCRIPTION:
Diabetes mellitus is one of the leading causes of illness worldwide. Diabetes can affect nerves, skin and blood vessels. Diabetics with problems in the patients nerves can lose the sense of touch in the patient's feet (called neuropathy) and so may unknowingly cause damage to the skin resulting in skin loss or an 'ulcer'. Diabetics also have difficulty healing any damaged tissues especially if the patient have diseased blood vessels causing a lack of blood to areas of the body including the feet (called ischaemia). Therefore diabetics have a greater chance of having an ulcer and a higher chance that it does not heal up. The loss of a protective skin barrier means that bacteria can enter the foot causing infections which can spread to bone and beyond. Ultimately this can result in gangrene, amputation or even death.

Stem or progenitor cells help repair and replace damage in the body. Blood vessels are key to this repair. Recent research has suggested that special progenitor cells found in the blood may be responsible. They are called Endothelial Progenitor Cells (EPCs) and seem to be in fewer numbers and are less effective at repair in diabetics.

Current treatments for diabetic wounds are not always successful and so the investigators need more research to look at new treatments. One possibility is to use electrical stimulation of nerves in the leg. Research studies have shown this may improve blood circulation and healing of wounds. This research will assess EPCs to see if they are linked to ulcer healing in diabetic patients with neuropathy only or with ischaemia as well. Furthermore the investigators wish to investigate whether electrical stimulation can affect progenitor cells and wound healing in these patients. The longterm goal of this research is to help diabetic patients improve their quality of life by reducing wound related complications

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients with Type 1 or 2 diabetes.
* Male or female, aged 18-85 years.
* Presence of significant neuropathic ulcers.
* Presence of significant neuroischaemic ulcers.
* Patients who are able and willing to follow the protocol requirements.

Exclusion Criteria:

* Unreliable, unwilling or unable to comprehend informed consent.
* Patients with recently diagnosed or with suspected deep vein thrombosis (DVT).
* Patients without neuroischaemic/ neuropathic ulcers
* Patients with cardiac demand pacemakers.
* Patients who are pregnant.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Improvement in ulcer size at monthly intervals up to 12 months follow up. | 12 months
  The wound will be measured after the electrical stimulation produced by Geko device is applied.

SECONDARY OUTCOMES:
Proportion of wounds healed at monthly intervals up to 12 months followup | 12 months
  Percentage of wounds healed after the electrical stimulation produced by Geko device is applied.